CLINICAL TRIAL: NCT05952622
Title: Comparison of Functional and Patient-reported Outcome Using Continuous Passive Motion in Rehabilitation After Plate Osteosynthesis of Proximal Humerus Fractures
Brief Title: Outcome After Plate Osteosynthesis of Proximal Humerus Fractures Using Continous Passive Motioning Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPM
Record Dates: First submitted 2023-04-19; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Proximal Humerus Fracture
Keywords: proximal humerus fracture; plate osteosynthesis; rehabilitation; continuous passive motion
MeSH Terms: interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Intervention Model Description: Patients are assigned to one of two rehabilitation protocols consisting of either A: initial immobilization followed by physiotherapy or B: initial immobilization followed by physiotherapy and additional continuous passive motion therapy
Masking Description: Patients are randomly assigend, masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehabilitation protocol (No Intervention): Standard rehabilitation after surgical treatment consisting of initial immobilization followed by physiotherapy.
- Rehabilitation protocol with CPM (Active Comparator): Additional treatment of patients with continuous passive motion after initial immobilization for 6 weeks.
  Interventions: Device: Continuous passive motion therapy

INTERVENTIONS:
Device: Continuous passive motion therapy — Patients will be supplied with a continuous passive motion device which will allow additional individual treatment of the affected shoulder for 6 weeks.
  Arms: Rehabilitation protocol with CPM

SUMMARY:
Patients suffering from a proximal humerus fracture treated with plate osteosynthesis will receive either regular aftercare (physiotherapy) or aftercare assisted with continous passive motion (physiotherapy + CPM). Change in functional and patient-reported outcome (PROM) over time will be evaluated and compared.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, monocentric study focusing on the rehabilitation process after surgical treatment of proximal humerus fractures. Patients treated with plate osteosynthesis and eligible to participate will be randomly assigend to either a regular rehabilitation protocol (immobilization and physiotherapy) or a rehabilitation protocol with the additional use of a continous passive motion device (immobilization, physiotherapy and CPM).

After 6 and 12 weeks as well as 1 year in a follow-up examination functional (range of motion) and patient-reported outcome (Disabilities of Arm, Shoulder and Hand Score [DASH], Constant-Score, pain on visual analogue scale, subjective satisfaction) will be evaluated. Results will be compared towards possible differences and effect of CPM therapy. In addition demographic factors (age, sex, BMI, etc.) and complications will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* patients with proximal humeral fracture treated with plate osteosynthesis during the enrollment period
* understanding of German language (written and oral)
* written informed consent of the patient or the legal guardian

Exclusion Criteria:

* patients not meeting the aforementioned criteria
* patients with the need of / or an already existing endoprosthesis
* patients with ipsilateral fracture of the distal radius
* patients with cerebral damage (contusio or commotio cerebri)
* patients with affection of the brachial plexus or nerve palsy
* non-compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Range of Motion (ROM) after 6 weeks, 12 weeks and 1 year | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Objetive functional clinical result. Evaluation ot Motion of the shoulder in ° measured via goniometer. Physiological Abduction/Adduction: 180/0/40°, Anteversion/Retroversion 160/0/40°, external/internal rotation: 70/0/60°
Change of Disabilities of Arm, Shoulder and Hand Score (DASH) after 6 weeks, 12 weeks and 1 year | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Evaluation of the subjective function (patient reported outcome) using the DASH-Score, 0-100, best: 0, worst: 100
Change of Constant-Score (CSS) after 6 weeks, 12 weeks and 1 year | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Evaluation of the subjective function (patient reported outcome) using the Constant-Score, 0-100, best: 100, worst: 0
Change of Pain on visual analogue scale (VAS) after 6 weeks, 12 weeks and 1 year | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Evaluation of the subjective pain using a visual analogue scale, 0-10, best:0, worst: 10
Change of Subjective satisfaction with surgical treatment (SSV) after 6 weeks, 12 weeks and 1 year | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Evaluation of the subjective satisfaction using the subjective shoulder value, 0-100, best:100, worst: 0

SECONDARY OUTCOMES:
Influence of demographic factors upon rehabilitation process | Time of Follow-Up assesment, 6 and 12weeks as well as 1year after surgical treatment
  Evaluation of the underlying demographic factors (gender, age, BMI) and whether these affect the functional and patient-reported outcome (univariate regressional analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden, TU Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tille E, Lorenz F, Beyer F, Schlussler A, Biewener A, Nowotny J. Early functional improvements using continuous passive motion therapy after angular-stable plate osteosynthesis of proximal humerus fractures - results of a prospective, randomized trial. J Orthop Surg Res. 2024 May 28;19(1):313. doi: 10.1186/s13018-024-04804-x. PMID 38802866